CLINICAL TRIAL: NCT05430932
Title: Effect Of Laparoscopic Sleeve Gastrectomy (LSG) on Vitamin D, Parathormone and Calcium Levels
Brief Title: Effect Of Laparoscopic Sleeve Gastrectomy on Vitamin D, Parathormone and Calcium Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Aouf, Dr, assistant lecturer of General Surgery, Kafrelsheikh University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKSU50-5-24
Record Dates: First submitted 2022-06-18; First posted 2022-06-24 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Vitamin D Deficiency; Calcium Deficiency
MeSH Terms: conditions — Obesity, Morbid; Vitamin D Deficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laparoscopic sleeve gastrectomy (Experimental): After sleeve gastrectomy, assessment of vitamin D, calcium and parathormone levels is performed.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Laparoscopic resection of a part of the stomach to enable the patient to lose weight.

SUMMARY:
Obesity is likely to be the disease of the 21th century. The growth of obesity is worldwide, a pandemic, and has increased globally in the last 30 years. Developed countries were more affected, but developing countries have increasingly contributed to this epidemic as they continue to modernize. The national and global burden of obesity, with its public health and financial implications, is projected to increase markedly in the next two decades.

the study aimed to assess the effect of Vit D supplementation on preventing altered levels of calcium, Vit D, and parathormone after laparoscopic sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* male or female
* from 18 to 60 ages
* BMI: 40 kg/m2 or > 35 kg/m2
* comorbidities e.g., hypertension and DM
* conservative management for obesity failed in at least 2 years

Exclusion Criteria:

* BMI > 60
* history of bariatric surgery
* symptomatic reflux oesophagitis
* stomach cancer
* active peptic ulcer disease
* alcohol or drug abuse
* major psychological disturbance
* major eating troubles
* risky anesthesia
* risky surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Vitamin D level assessment | 1 year
  Assessment of the vitamin D level after sleeve gastrectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafr el-Sheikh Governorate, Egypt